CLINICAL TRIAL: NCT02725320
Title: Rotator Cuff Surgical Outcomes in Women
Acronym: RCSOW
Status: Unknown | Type: Observational
Last Known Status: Active, not recruiting
Sponsor: University of Calgary (Other)
Responsible Party: Principal Investigator, Marlis Sabo, Clinical Assistant Professor, University of Calgary
Other Study IDs: REB15-1229
Record Dates: First submitted 2016-03-03; First posted 2016-03-31 (Estimated); Last update posted 2019-04-26 (Actual); Status verified 2019-04

CONDITIONS: Injury of Shoulder Region; Rotator Cuff Syndrome
Keywords: rotator cuff; shoulder reconstruction
MeSH Terms: conditions — Shoulder Injuries

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- Female Rotator Cuff Surgical Group: Females, 35-75 receiving surgery for predominantly unilateral rotator cuff syndrome
- Male Rotator Cuff Surgical Group: Males, 35-75 receiving surgery for predominantly unilateral rotator cuff syndrome

SUMMARY:
The overall purpose of this work is to use a prospective cohort study to examine patient-specific but shoulder-extrinsic factors and how they influence the results of rotator cuff surgery. There are undoubtedly many factors that play a role in patient outcome, however, this project will focus on three: the effect of gender on outcome, the effect of mood disorders and coping style on outcome, and the effect of patient height and reach on outcome after rotator cuff surgery. It is hypothesized that these factors will have a significant influence over outcomes.

ELIGIBILITY:
Inclusion Criteria:

* Referred for surgical treatment of predominantly unilateral rotator cuff syndrome

Exclusion Criteria:

* unable to speak or read English
* unable to complete 12 month follow-up
* significant cervicogenic arm and shoulder pain in the affected arm
* significant chronic pain diagnoses felt at least as likely to be the cause of the symptoms as the rotator cuff condition as evaluated by the surgeon

Ages: 35 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The participants for this study will be selected from the practice of three shoulder reconstruction surgeons in their embedded clinical research practice.
Sampling Method: Non-Probability Sample
Enrollment: 192 (Actual)
Dates: Start 2016-02; Primary Completion 2020-12 (Estimated); Study Completion 2020-12 (Estimated)

PRIMARY OUTCOMES:
Western Ontario Rotator Cuff score (WORC) | 1 year
  WORC scores will be compared at 12 months between the groups (males versus females)

SECONDARY OUTCOMES:
Overall change in WORC (male versus female) | 1 year
  Evaluation of the overall change in WORC score by gender
Rate of change in WORC (male versus female) | 1 year
  Evaluation of the rate of change in WORC score over 1 year between male and female
Rate of change in visual analogue scale (VAS) (male versus female) | 1 year
  Evaluation of the rate of change in VAS score over 1 year between male and female
Rate of change in SF-36 (short-form 36) response scores (male versus female) | 1 year
  Evaluation of the rate of change in SF-36 scores over 1 year between male and female
Rate of change of satisfaction with surgical outcome (male versus female) | 1 year
  Evaluation of the rate of change in satisfaction with surgical outcome between male and female over 1 year
Prevalence of anxiety and depression at baseline | Baseline data
  Evaluation of the HADS (Hospital Anxiety and Depression Scale) at baseline to determine the prevalence of mood disorder
Prevalence of catastrophizing at baseline | Baseline data
  Evaluation of the PCS (Pain Catastrophizing Score) at baseline to determine the prevalence catastrophizing
Improvement in HADS | 1 year
  Evaluation of HADS scores over 1 year to determine improvement from baseline
Height (males versus females) | baseline
  Evaluation of the difference in height between genders
Change in reach over time | 1 year
  Evaluation of forward reach to determine the change from baseline to one year
WORC score by HADS score | 1 year
WORC score by PCS score | 1 year
WORC score by forward reach | 1 year
WORC score correlated to gender, PCS, HADS | 1 year

CONTACTS AND LOCATIONS:
Overall Officials: Marlis Sabo, MD, FRCSC, Principal Investigator — University of Calgary
Locations (1):
- South Health Campus, Calgary, Alberta, Canada

IPD SHARING:
Plan to Share IPD: No